CLINICAL TRIAL: NCT01072318
Title: Evaluate Efficacy and Safety of Extended Adjuvant Treatment With Letrozole in Postmenopausal Women With Hormone Receptor Positive Breast Cancer Who Have Completed 5 Years of Toremifene
Brief Title: Extended Adjuvant Treatment With Letrozole in Breast Cancer Who Complete 5 Years of Toremifene
Acronym: LEXTOP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Korean Breast Cancer Study Group (Other)
Responsible Party: Sei-Hyun Ahn, Asan medical center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBCSG007
Record Dates: First submitted 2010-02-14; First posted 2010-02-22 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; extended adjuvant hormonal therapy; letrozole; Toremifene
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Letrozole, DFS (Experimental): Efficacy evaluation of extended letrozole after 5 year fareston use
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5mg
  Other Names: Femara

SUMMARY:
The purpose of this study is to assess Efficacy and Safety of Extended Adjuvant Treatment With Letrozole in Postmenopausal Women With Hormone Receptor Positive Breast Cancer Who Complete 5 Years of Toremifene

DETAILED DESCRIPTION:
1. Primary purpose To evaluate disease free survival rate (DFS) after taking 36 months with Letrozole in postmenopausal women with hormone receptor positive breast cancer who complete 5 years of Toremifene
2. Secondary purpose

   * To evaluate follows after taking 36 months with Letrozole in postmenopausal women with hormone receptor positive breast cancer who complete 5 years of Toremifene.

     1. Disease Free Survival rate(DFS)-12 months, 24 months
     2. Distant disease free survival rate(DDFS), Overall Survival(OS)
   * 12 months, 24 months, 36 months c. safety
   * Change of lipid profiles
   * Mortality and morbidity due to Cardiovascular disease
   * Incidence of Fracture
   * Change of Bone density
   * Common toxic effect

ELIGIBILITY:
Inclusion Criteria:

1. Patients have undergone surgery of the breast cancer and proven histologically to be invasive breast cancer.
2. Removed the breast cancer histologically or cytologically
3. No evidence of breast cancer in controlateral breast
4. No evidence of metastasis
5. Postmenopausal Women With Hormone Receptor Positive Breast Cancer Who Complete 5 Years of Toremifene in 30 months
6. Postmenopausal state was defined the following conditions, at least one of a, b

   1. Serum FSH ≥ 30 mIU/mL
   2. Amenorrhea ≥ 1 year
7. Estrogen receptor(+) or Progesterone receptor(+)
8. No Evidence of Recurrence

Exclusion Criteria:

1. Patient with hormone receptor negative
2. Patients with malignancies
3. Patients with other aromatase inhibitor and chemotherapy
4. Patients with Other hormone therapy and Hormonal replacement therapy
5. Patients with Hormone replacement therapy during taking Toremifene
6. Estimated life expectancy of <12 months
7. WBC<3,000/mm3 or Platelet count<100,000/mm3
8. AST and/or ALT ≥2xUNL
9. Alkaline phosphatase ≥2xUNL

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival rate | 3 years

SECONDARY OUTCOMES:
Disease free survival rate | 12 months, 24 months
Distant disease free survival rate | 12 months, 24 months, 36 months
Overall survival rate | 12, 24, 36 months
Toxicity was assessed by NCI-CTC version 3.0 | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Sei-Hyun Ahn, MD, Principal Investigator — Department of Surgery, Asan medical center, South Korea
Locations (1):
- Department of Surgery, Asan medical center, Seoul, South Korea